CLINICAL TRIAL: NCT02253758
Title: Arousal Pathways and Emergence From Sedation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Dr. Michal Roll, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TASMC-14-IM-0383-CTIL
Record Dates: First submitted 2014-08-10; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Anesthesia
Keywords: Magnetic Resonance Imaging; Electroencephalography; Conscious Sedation; Deep Sedation; Arousal; Consciousness
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sedation (Experimental): Volunteers will be sedated to Ramsay score 4-5 with propofol, and data will be recorded during arousal
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol will be injected as a continuous infusion by TCI intravenously
  Other Names: Propofol Liporum 1%

SUMMARY:
Emergence from sedation involves an increase in both the level of consciousness and arousal. Some insight to the neural core of consciousness was gained in the recent past. Our research objective is to characterize for the first time the spatiotemporal mobilization of the ascending reticular activating system during emergence from sedation; stated otherwise - to capture the neural core of arousal.

To achieve this objective we plan to utilize the advanced imaging modality of EEG-fMRI. In short, volunteers will be placed in the MRI. Following baseline recordings they will be sedated with a continuous drip of propofol, titrated to deep sedation. Once in that sedation level, propofol administration will cease until emerging to an awake-calm/light sedation.

Continuous EEG recordings and fMRI scans will be taken, both task specific (auditory oddball) and resting-fMRI. Analyses will focus (but will not be restricted to) on constituents of the ascending reticular activating system.

The expected advances of this proposal are:

1. Emergence from sedation (and anesthesia) is one of the critical stages and least elucidated area in the practice of anesthesia. Delayed awakening of varying degree is not uncommon after anesthesia and may have a number of different causes, individual or combined, which may be both drug or non-drug related, thus causing a diagnostic dilemma. Eventually - better insight into this subject will lead to better clinical practice and better understanding why patients emerge in such a diverse and sometimes unexpected manner.
2. Knowledge of the internal structure underlying arousal from anesthesia will help develop / upgrade brain monitors that could tell the anesthesiologist the patient's level of consciousness and prediction of arousal.
3. A detailed reproducible mapping of the arousal process may serve as the core of a drug screening platform for drugs that may expedite patient arousal.
4. Elucidation of the arousal paradigm from sedation will enhance our knowledge of physiological sleep.

Research hypothesis

Return of consciousness is a complex phenomenon comprising of interplay between the cortex and deeper brain structures. We hypothesize that the activation signature is conserved and similar between subjects. Furthermore, we hypothesize that inter-subject variability will arise mainly in the time domain, as evident from the clinical observation of variable time to emergence in different patients.

DETAILED DESCRIPTION:
Sedation and general anesthesia are at the hub of modern medicine. The practice of the administration of anesthesia and sedation has evolved considerably and is now considered safe and reproducible. Still, one of the critical parts of anesthesia practice is the emergence: with the phenomenological variability of the clinical presentations of emergence, and its increased inherent risks of airway patency, insufficient respiratory mechanics, hyperreflexia and altered mental state.

Our understanding of the underlying mechanisms of sedation and anesthesia is still somewhat lacking: The body of evidence concerning induction and maintenance is more evolved[1-4], whereas the most profound gaps of knowledge concern emergence.

While anesthetic agent exert a global effect on the brain, it is clear that some foci are more sensitive[5] and more relevant to the achievement of the anesthetic goals of hypnosis, amnesia, and reduced responsiveness.

Mechanisms of unconsciousness induced by general anesthesia[1] can be broadly dissected to two elements: consciousness and arousal: Current consciousness theories[6,7] ascribe to consciousness the ability to experience. To achieve that goal, information complexity and information integration are paramount. These faculties reside mainly in the neocortex. Arousal on the other hand, resides mainly in the thalamus, hypothalamus, midbrain and pons with the neural machinery of physiological sleep[8,9]. We tend to associate consciousness with arousability. Dreaming however - is a straightforward example of consciousness without arousal.

A given level of arousal is the output of the balance of the mutual inhibition between the sleep promoting locus - the ventrolateral preoptic nucleus - and the multiple arousal loci, commonly known as the ARAS (Ascending Reticular Activating System)[10,11]. Shortly, this dispersed system is comprised of multiple nuclei with different neurotransmitters. Some of the nuclei have thalamic projections and some are extra-thalamic with direct and diverse cortical projections. The transition between sleep and wakefulness is further enhanced by the Orexigenic neurons in the hypothalamus[12,13], which serve as a flip flop mechanism.

The research into consciousness has made some progress[14] using anesthetic approaches and most specifically, emergence from sedation and anesthesia, to describe the neural core of consciousness. Recently, publications by Purdon et al.[15,16] identified an EEG signature of consciousness transition state.

The body of evidence concerning arousal pathways is less formidable, possibly due to the dispersed array of nuclei, and their "deep" subcortical locations, complicating their evaluation in less invasive methods (such as scalp EEG). The classic research tool of this field is lesions studies (both in animal models and unfortunate patients)[17,18] in discrete loci with an observed change in sleep-wake physiology. Recently, pioneering ex vivo (rat pups midbrain slices) research by Garcia-rill and Charlesworth[19], using intracellular recordings provided compelling data supporting electrical coupling and coherence of neurons within nuclei of the ARAS. However, to the best of our knowledge to this date there has been no explicit trial to capture or characterize the dynamic changes in the ARAS of human subjects emerging from sedation.

Research objectives

1. To characterize the spatiotemporal signature sequence of the arousing brain, focusing (but not restricted to) on deep brain structures. Arousal signature may include the following:

   * A conserved sequence of brain structures mobilization.
   * Summation of foci activations (without an explicit order).
   * Hierarchy between different loci (cholinergic vs. monoaminic components of the ARAS).
2. To identify a reproducible signal heralding imminent return of consciousness.

Methods:

The proposed study has been submitted to the Institutional Review Board committee for approval.

Experiment summary:

The proposed study is an interventional, single center study, conducted on 20 volunteers. A sample size of 20 was chosen in light of the relatively low signal to noise ratio inherent to fMRI imaging. subjects will be healthy males age 20-40, who are not taking chronic medications or using illicit drugs. All subjects, after signing the informed consent form, will fill a standard MRI questionnaire for the detection of metallic implants and will undergo medical evaluation and examination by the anesthesiologist. During the study period volunteers will be monitored by non invasive standard patient ASA monitoring: ECG, blood pressure, pulse oximetry, and exhaled CO2 levels. Each subject will be connected to an EEG recording cap, and will be placed in the magnet. Baseline recordings of EEG, MRI and fMRI will be taken. Then sedation will be induced with continuous IV propofol infusion with a Target Controlled Infusion pump - TCI, using the Marsh model[14,20,21]. Depth of sedation will be titrated to deep sedation (Ramsay scale 5)[22]. Subsequently, propofol administration will be discontinued, and continuous EEG and fMRI recordings will be taken until emerging from sedation to an awake calm/light sedation (Ramsay 2-3), as verified by a response to the subject's given name. At this point EEG monitoring and fMRI scans will cease. The subject will be helped out of the magnet and transferred to a post anesthesia care unit (PACU).

All subjects will be monitored until reaching discharge criteria ascertained by an examination performed by an anesthesiologist.

Brain monitoring

1. Functional Magnetic Resonance (fMRI): brain BOLD fMRI - blood oxygen level dependent fMRI - harnessing the magnetic properties of the ferric ion of hemoglobin to image changes in blood flow to metabolically active brain loci. The underlying assumption of the imaging modality (similar to Positron Emission Tomography) is the metabolic coupling of cellular activity and blood flow. Analyses will focus but will not be restricted to subthalamic structures involved in the RAS.
2. EEG (electroencephalogram), while in the MRI - EEG-fMRI. Combining the superior temporal resolution of the EEG with the localizing resolution of the MRI. The EEG will serve as an adjunct to the level of sedation and as source for data concerning thalamocortical pathways or arousal.

Expected results:

The results from this research project may help improve patient safety through the prediction of his/her arousal status. Anesthesia/Arousal level monitors have yet to prove their contribution to patient safety. Integration of deep brain structures data may prove to be the missing link to improving monitors' performance. Additionally, a thorough understanding of the arousal process can potentially help develop agents to hasten arousal, as it may serve as a screening paradigm for known pharmaceuticals (expanding their clinical indications) as well as new chemical entities (NCEs).

Feasibility and perceived strengths:

The feasibility of the proposed research project is very high. The project will be performed in Tel Aviv Medical Center in the Wohl Center for Advanced Imaging. The Wohl Center involves a prominent neuroscience research group with a significant number of publications related to emotional and cognitive processing in health and disease. Some of these studies include volunteers[23,24] and the use of fMRI and EEG to follow propofol induced sedation[25,26]. The proposed project will enjoy a full collaboration with the research center. In this light, the completion of the proposed imaging sessions and their subsequent analyses is realistic.

A thorough characterization of the emergence process warrants careful, dedicated attention to deep brain structures while designing the experiment throughout its execution and during analyses. As stand-alone scalp EEG recordings have fallen short of finding the "emergence fingerprint" (as EEG signal represent mostly cortical activity) we contest that a combined EEG-fMRI carries more hopes for the characterization of emergence from sedation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males (ASA scale 1-2), volunteers only

Exclusion Criteria:

* Use of chronic medications or illicit drugs
* Metallic implants
* Previous brain injury
* General anaesthesia up to a week earlier to research examination
* Known drug sensitivity to Propofol, soybean oil or peanuts

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of brain network connectivity underlying arousal from anesthesia. | Data collection time frame will not exceed one hour post propofol infusion cessation.
  Network connectivity of brain loci involved in arousal pathways will be evaluated for each patient at these time points: baseline, deep sedation and return to conscious state. The identification of these time points will be decided according to the Ramsay clinical scale for sedation depth. A score of 2 for baseline, 5 for deep sedation, and 2-3 for regaining consciousness. An external validation for these time points will derive from the oddball auditory test, in which the brain reaction to a sound in a different pitch is recorded. In the sedated state this reaction is perturbed.

SECONDARY OUTCOMES:
Characterization of the internal structure and temporal hierarchy underlying arousal from anesthesia. | Data collection time frame will not exceed one hour post propofol infusion cessation.
  At the group level an attempt will be made to discern temporal hierarchy (which of the aforementioned nuclei is the first to regain activity within the network) between the different ROIs (in voxels and normalized to a standarized brain) involved in the arousal pathways. The basal forebrain, laterodorsal tegmental nuclei, pedunculupontine nuclei, the ventral hypothalamus and the thalamus will all be included in the putative connectivity map.

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, Prof. M.D., Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Division of Anesthesia, Pain and Critical Care, Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Whol Institute for Advanced Imaging, Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Lee U, Mashour GA, Kim S, Noh GJ, Choi BM. Propofol induction reduces the capacity for neural information integration: implications for the mechanism of consciousness and general anesthesia. Conscious Cogn. 2009 Mar;18(1):56-64. doi: 10.1016/j.concog.2008.10.005. Epub 2008 Dec 2. PMID 19054696
- [Background] Breshears JD, Roland JL, Sharma M, Gaona CM, Freudenburg ZV, Tempelhoff R, Avidan MS, Leuthardt EC. Stable and dynamic cortical electrophysiology of induction and emergence with propofol anesthesia. Proc Natl Acad Sci U S A. 2010 Dec 7;107(49):21170-5. doi: 10.1073/pnas.1011949107. Epub 2010 Nov 15. PMID 21078987
- [Background] Hwang E, Kim S, Han K, Choi JH. Characterization of phase transition in the thalamocortical system during anesthesia-induced loss of consciousness. PLoS One. 2012;7(12):e50580. doi: 10.1371/journal.pone.0050580. Epub 2012 Dec 7. PMID 23236379
- [Background] Alkire MT, Hudetz AG, Tononi G. Consciousness and anesthesia. Science. 2008 Nov 7;322(5903):876-80. doi: 10.1126/science.1149213. PMID 18988836
- [Background] Tononi G. An information integration theory of consciousness. BMC Neurosci. 2004 Nov 2;5:42. doi: 10.1186/1471-2202-5-42. PMID 15522121
- [Background] Tononi G, Koch C. The neural correlates of consciousness: an update. Ann N Y Acad Sci. 2008 Mar;1124:239-61. doi: 10.1196/annals.1440.004. PMID 18400934
- [Background] Franks NP. General anaesthesia: from molecular targets to neuronal pathways of sleep and arousal. Nat Rev Neurosci. 2008 May;9(5):370-86. doi: 10.1038/nrn2372. PMID 18425091
- [Background] Brown EN, Purdon PL, Van Dort CJ. General anesthesia and altered states of arousal: a systems neuroscience analysis. Annu Rev Neurosci. 2011;34:601-28. doi: 10.1146/annurev-neuro-060909-153200. PMID 21513454
- [Background] Saper CB, Chou TC, Scammell TE. The sleep switch: hypothalamic control of sleep and wakefulness. Trends Neurosci. 2001 Dec;24(12):726-31. doi: 10.1016/s0166-2236(00)02002-6. PMID 11718878
- [Background] Solt K. General anesthesia: activating a sleep switch? Curr Biol. 2012 Nov 6;22(21):R918-9. doi: 10.1016/j.cub.2012.09.033. PMID 23137688
- [Background] Baumann CR, Bassetti CL. Hypocretins (orexins) and sleep-wake disorders. Lancet Neurol. 2005 Oct;4(10):673-82. doi: 10.1016/S1474-4422(05)70196-4. PMID 16168936
- [Background] Kelz MB, Sun Y, Chen J, Cheng Meng Q, Moore JT, Veasey SC, Dixon S, Thornton M, Funato H, Yanagisawa M. An essential role for orexins in emergence from general anesthesia. Proc Natl Acad Sci U S A. 2008 Jan 29;105(4):1309-14. doi: 10.1073/pnas.0707146105. Epub 2008 Jan 14. PMID 18195361
- [Background] Langsjo JW, Alkire MT, Kaskinoro K, Hayama H, Maksimow A, Kaisti KK, Aalto S, Aantaa R, Jaaskelainen SK, Revonsuo A, Scheinin H. Returning from oblivion: imaging the neural core of consciousness. J Neurosci. 2012 Apr 4;32(14):4935-43. doi: 10.1523/JNEUROSCI.4962-11.2012. PMID 22492049
- [Background] Mukamel EA, Pirondini E, Babadi B, Wong KF, Pierce ET, Harrell PG, Walsh JL, Salazar-Gomez AF, Cash SS, Eskandar EN, Weiner VS, Brown EN, Purdon PL. A transition in brain state during propofol-induced unconsciousness. J Neurosci. 2014 Jan 15;34(3):839-45. doi: 10.1523/JNEUROSCI.5813-12.2014. PMID 24431442
- [Background] Purdon PL, Pierce ET, Mukamel EA, Prerau MJ, Walsh JL, Wong KF, Salazar-Gomez AF, Harrell PG, Sampson AL, Cimenser A, Ching S, Kopell NJ, Tavares-Stoeckel C, Habeeb K, Merhar R, Brown EN. Electroencephalogram signatures of loss and recovery of consciousness from propofol. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):E1142-51. doi: 10.1073/pnas.1221180110. Epub 2013 Mar 4. PMID 23487781
- [Background] Moruzzi G, Magoun HW. Brain stem reticular formation and activation of the EEG. Electroencephalogr Clin Neurophysiol. 1949 Nov;1(4):455-73. PMID 18421835
- [Background] Schmidt C, Collette F, Leclercq Y, Sterpenich V, Vandewalle G, Berthomier P, Berthomier C, Phillips C, Tinguely G, Darsaud A, Gais S, Schabus M, Desseilles M, Dang-Vu TT, Salmon E, Balteau E, Degueldre C, Luxen A, Maquet P, Cajochen C, Peigneux P. Homeostatic sleep pressure and responses to sustained attention in the suprachiasmatic area. Science. 2009 Apr 24;324(5926):516-9. doi: 10.1126/science.1167337. PMID 19390047
- [Background] Garcia-Rill E, Kezunovic N, Hyde J, Simon C, Beck P, Urbano FJ. Coherence and frequency in the reticular activating system (RAS). Sleep Med Rev. 2013 Jun;17(3):227-38. doi: 10.1016/j.smrv.2012.06.002. Epub 2012 Oct 6. PMID 23044219
- [Background] Schroter MS, Spoormaker VI, Schorer A, Wohlschlager A, Czisch M, Kochs EF, Zimmer C, Hemmer B, Schneider G, Jordan D, Ilg R. Spatiotemporal reconfiguration of large-scale brain functional networks during propofol-induced loss of consciousness. J Neurosci. 2012 Sep 12;32(37):12832-40. doi: 10.1523/JNEUROSCI.6046-11.2012. PMID 22973006
- [Background] Marsh B, White M, Morton N, Kenny GN. Pharmacokinetic model driven infusion of propofol in children. Br J Anaesth. 1991 Jul;67(1):41-8. doi: 10.1093/bja/67.1.41. PMID 1859758
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Meir-Hasson Y, Kinreich S, Podlipsky I, Hendler T, Intrator N. An EEG Finger-Print of fMRI deep regional activation. Neuroimage. 2014 Nov 15;102 Pt 1:128-41. doi: 10.1016/j.neuroimage.2013.11.004. Epub 2013 Nov 15. PMID 24246494
- [Background] Abraham E, Hendler T, Shapira-Lichter I, Kanat-Maymon Y, Zagoory-Sharon O, Feldman R. Father's brain is sensitive to childcare experiences. Proc Natl Acad Sci U S A. 2014 Jul 8;111(27):9792-7. doi: 10.1073/pnas.1402569111. Epub 2014 May 27. PMID 24912146
- [Background] Weinstein M, Ben-Sira L, Levy Y, Zachor DA, Ben Itzhak E, Artzi M, Tarrasch R, Eksteine PM, Hendler T, Ben Bashat D. Abnormal white matter integrity in young children with autism. Hum Brain Mapp. 2011 Apr;32(4):534-43. doi: 10.1002/hbm.21042. PMID 21391246
- [Background] Ben Bashat D, Kronfeld-Duenias V, Zachor DA, Ekstein PM, Hendler T, Tarrasch R, Even A, Levy Y, Ben Sira L. Accelerated maturation of white matter in young children with autism: a high b value DWI study. Neuroimage. 2007 Aug 1;37(1):40-7. doi: 10.1016/j.neuroimage.2007.04.060. Epub 2007 May 18. PMID 17566764